CLINICAL TRIAL: NCT04554394
Title: A Prospective, Non-Randomized, Multicenter Pivotal Study of Nano-Pulse Stimulation™ (NPS™) Treatment of Cutaneous Non-Genital Warts
Brief Title: CellFX System for the Treatment of Cutaneous Non-Genital Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-WP-010
Record Dates: First submitted 2020-08-29; First posted 2020-09-18 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Warts; Warts Hand; Verruca
Keywords: CellFX; Nano-Pulse Stimulation; NPS; Clearance
MeSH Terms: conditions — Warts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CellFX Treated Wart (Experimental): Treated wart with CellFX device intervention
  Interventions: Device: CellFX Device
- Non-treated Wart (No Intervention): Control wart for each enrolled subject without intervention

INTERVENTIONS:
Device: CellFX Device — The CellFX System utilizes non-thermal, localized delivery of a timed series of low energy, nanosecond electrical pulses that can trigger regulated cell death.
  Arms: CellFX Treated Wart

SUMMARY:
This prospective, non-randomized, multicenter pivotal study is designed to evaluate the safety and effectiveness of the CellFX System in patients with cutaneous non-genital warts on all areas of the body, excluding the face.

DETAILED DESCRIPTION:
The study will enroll healthy adult subjects with a minimum of two cutaneous non-genital warts, excluding the face, with each wart lesion not exceeding 10 x 10mm. One of the warts for each subject will be untreated and will serve as the subject's internal control. Macrophotography of all study warts will be captured along with Investigator assessments using the Wart Measurement Scale (WMS) and lesion measurements for wart reduction. All subjects will be followed at 7, 30, 60, 90 and 120-days post-initial CellFX treatment. All wart lesions are eligible for re-treatment up to 3 times over the course of the study. Adverse events will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 21 and not older than 80 years of age
* Subjects must be able to read and speak English or Spanish
* Subjects must sign a written informed consent to participate in the study, prior to any study related procedures
* Subject must have a minimum of two cutaneous non-genital warts, each not exceeding 10 x 10mm
* Subject is willing to undergo all study-mandated procedures
* Subject agrees to refrain from using all other wart removal products or treatments (topical medication including over-the-counter medications) during the study period

Exclusion Criteria:

* Subject has an implantable electronic medical device. (pacemaker, implantable cardioverter defibrillator, etc.)
* Subject has cochlear implants
* Subject has an active systemic infection or history of an infection in the designated treatment area within 90 days of enrollment
* Subject has a history of and/or current tinnitus
* Subject is known to be immune-compromised
* Subject is taking a blood thinning medication (Antiplatelet, Anticoagulation, Factor Xa Inhibitor, etc.)
* Subject has Type 1 Diabetes and is insulin dependent
* Subject has a known allergy to Lidocaine or Lidocaine-like products
* Subject is a member of a vulnerable population including individuals employed by the Sponsor, clinic site, or entity associated with the conduct of the study
* Subject has a comorbidity or condition which may reduce compliance with this protocol, including follow-up visits
* Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nuccitelli, PhD, Study Chair — Pulse Biosciences, Inc.
Locations (5):
- United States (5):
  - Investigate MD, LLC, Scottsdale, Arizona
  - Scripps Clinic Carmel Valley, San Diego, California
  - Skin Search of Rochester, Inc., Rochester, New York
  - Dermatology, Laser & Vein Specialists of the Carolinas, PLLC, Charlotte, North Carolina
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 62 study subjects were enrolled. A total of 257 warts were studied, including 195 warts assigned to treatment and 62 assigned to control arm.
Pre-assignment Details: 62 subjects were enrolled. One wart per subject was randomized and pre-assigned as the control.
Units Other Than Participants: lesions
Groups:
- CellFX Treated Warts: CellFX device using pre-defined energy protocols
  CellFX Device: The CellFX System utilizes non-thermal, localized delivery of a timed series of low energy, nanosecond electrical pulses that can trigger regulated cell death.
- Non-Treated Controls: Non-treated wart arm, one study wart per enrolled subject.
Period: Overall Study
Arm/Group | CellFX Treated Warts | Non-Treated Controls
Started | 62; 195 lesions | 62; 62 lesions (A total of 62 participants were enrolled and 1 randomized control wart per participant was enrolled in the control arm)
Completed | 53; 136 lesions | 53; 53 lesions
Not Completed | 9; 59 lesions | 9; 9 lesions
Not completed — Clinical Site Closed due to COVID-19 Restrictions | 4 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Subjects diagnosed with cutaneous warts, including common, flat and plantar subgroups
Groups:
- CellFX Treated Verrucae: CellFX device using pre-defined energy protocols
  CellFX Device: The CellFX System utilizes non-thermal, localized delivery of a timed series of low energy, nanosecond electrical pulses that can trigger regulated cell death.
Arm/Group | CellFX Treated Verrucae
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.3 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 58
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick skin phototypes (FSP) were developed in Boston in 1975 for use with phototherapy. The scale's original purpose was to help determine a patient's risk of burning or tanning when exposed to UV light. The current scale classifies skin from types I to VI. Type I refers to skin that always burns, while type VI refers to skin that never burns. In general, a lower FSP means a person's skin burns more easily than it tans. A higher FSP means that a person's skin does not burn easily.
  Participants
    Class I | 3
    Class II | 27
    Class III | 20
    Class IV | 12
Verrucae Disposition [Number; unit: warts]
  Treated | 195
  Control | 62
  Not treated | 10
Wart Subtype [Number; unit: warts] — Subtype of wart treated in the study
  warts
    Common | 195
    Plantar | 55
    Flat | 17
Anatomic Location [Number; unit: warts] — Location of wart lesion
  warts
    Hand | 131
    Foot | 79
    Leg | 23
    Knee | 10
    Ankle | 6
    Arm | 4
    Elbow | 3
    Wrist | 3
    Torso | 2
History of Prior Verrucae Treatment [Number; unit: warts]
  Cryotherapy | 49
  Over the Counter Medical Treatment | 40
  Laser Treatment | 10
  Over the Counter and Laser Treatment | 8
  Electrocautery | 7
  Cantharone and Cryotherapy | 4
  Investigational Product | 2
  Aldara and Cryotherapy | 1
  Laser Treatment and Cryotherapy | 1
  Yeast Injection | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Verrucae Cleared
Description: Percentage of Verrucae with Clearance (91-100% reduction)
Time Frame: 60-days post-last CellFX treatment
Population: Percent of verrucae clearance observed at 60-days post-last treatment. Reduction in verrucae size and/or clearance not assessed in the "Non-treated Control" Arm/Group or similar.
Measure: Number; unit: percentage of verrucae clearance
Units Other Than Participants: common verrucae
Groups:
- Warts Treated With CellFX (Common, Flat, and Plantar): CellFX device using pre-defined energy protocols
  CellFX Device: The CellFX System utilizes non-thermal, localized delivery of a timed series of low energy, nanosecond electrical pulses that can trigger regulated cell death.
Arm/Group | Warts Treated With CellFX (Common, Flat, and Plantar)
Number analyzed (Participants) | 53
Number analyzed (common verrucae) | 136
percentage of verrucae clearance | 67.6

2. Secondary Outcome: Subject Satisfaction
Description: Satisfaction with reduction in verrucae size or clearance of verrucae measured using the following scale; 5 (Satisfied), 4 (Mostly Satisfied), 3 (Partially Satisfied), 2 (Dissatisfied), 1 (Highly Dissatisfied)
Time Frame: 60-days post-last CellFX treatment
Population: All Treated Verrucae observed at 60-days post-last CellFX treatment
Measure: Number; unit: percentage of participants
Units Other Than Participants: total treated warts
Arm/Group | CellFX Treated Verrucae
Number analyzed (Participants) | 98
Number analyzed (total treated warts) | 133
percentage of participants | 73.7

ADVERSE EVENTS:
Time Frame: 4 months after initial CellFX Treatment
Groups:
- CellFX Treated Wart Lesion: CellFX device using pre-defined energy protocols
  CellFX Device: The CellFX System utilizes non-thermal, localized delivery of a timed series of low energy, nanosecond electrical pulses that can trigger regulated cell death.
Arm/Group | CellFX Treated Wart Lesion
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 8/62
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CellFX Treated Wart Lesion (N=62)
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 (3) — Transient Numbness at the Target Site resolving without medical intervention.
Pain (General disorders) | 2 (2) — Pain at Treatment Site treated with Motrin.
Infection (Infections and infestations) | 3 (3) — Suspect infection. Neosporin used in one subject and antibiotic used in second subject with both events resolving within 2 weeks. No cultures performed for both subjects. Third subject had a negative culture and event resolved within 5 days.
Numbness and swelling (General disorders) | 1 (1) — Numbness and swelling reported at the index finger of right hand and took Motrin as needed with resolution of event by 1-month.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT04554394/Prot_000.pdf